CLINICAL TRIAL: NCT00967746
Title: A Randomized, Multicenter, Explorative Trial to Explore the Safety, Acceptability and Vaginal Bleeding Pattern of Three Doses of an Etonogestrel-releasing Medicated Intrauterine System (ENG-MIUS) Versus a Copper-releasing Intrauterine Device (IUD)
Brief Title: An Explorative Trial to Explore the Safety, Acceptability and Vaginal Bleeding Pattern of Three Etonogestrel-releasing Medicated Intrauterine Systems (Study P06060)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P06060
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- ENG-MIUS low (Experimental): Low dose: ENG-MIUS containing 38 mg ENG with a skin thickness of approximately 350 μm
  Interventions: Drug: Etonogestrel-releasing IUS
- ENG-MIUS intermediate (Experimental): Intermediate dose: ENG-MIUS containing 61 mg ENG with a skin thickness of approximately 140 μm
  Interventions: Drug: Etonogestrel-releasing IUS
- ENG-MIUS high (Experimental): High dose: ENG-MIUS containing 72 mg ENG with a skin thickness of approximately 50 μm
  Interventions: Drug: Etonogestrel-releasing IUS
- Multiload (Active Comparator): Multiload-cu 375®
  Interventions: Device: Multiload-cu 375®

INTERVENTIONS:
Drug: Etonogestrel-releasing IUS — Low dose; treatment duration of 6 months with a possible extension to 12 months
  Other Names: SCH 900342; ORG 299001
  Arms: ENG-MIUS low
Drug: Etonogestrel-releasing IUS — Intermediate dose; treatment duration of 6 months with a possible extension to 12 months
  Other Names: SCH 900342; ORG 299001
  Arms: ENG-MIUS intermediate
Drug: Etonogestrel-releasing IUS — High dose; treatment duration of 6 months with a possible extension to 12 months
  Other Names: SCH 900342; ORG 299001
  Arms: ENG-MIUS high
Device: Multiload-cu 375® — Duration of 6 months with a possible extension to 12 months
  Arms: Multiload

SUMMARY:
This is a phase 2, randomized, active-controlled, parallel-group, multicenter, single-blind trial of three different doses of etonogestrel releasing medicated intrauterine systems (ENG-MIUS) in healthy parous women in need for contraception.

The primary trial objective is to explore safety and acceptability of three doses of an ENG-releasing medicated intrauterine system (ENG-MIUS) as compared to Multiload-cu 375®.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects in need for contraception will be selected to participate in the trial;
* Each subject must be >=18 to <=40 years of age at screening and in need for contraception;
* Each subject must have given birth to at least one child (gestational age >=28 weeks);
* Each subject must have a uterus with a measured length between 6.0 and 9.0 cm (extremes included) from external os to fundus uteri.

Exclusion Criteria:

* A subject must not be pregnant or suspected to be pregnant;
* A subject must not have had an ectopic pregnancy in the past or must not have a history or presence of predisposing factors for this condition such as salpingitis, endometritis or pelvic peritonitis;
* A subject must not have a history or presence of any malignancy;
* A subject must not have a history or presence of premalignant disease of the uterus or cervix, including endometrial hyperplasia, or (other) sex-steroid sensitive premalignancies;
* A subject must not have an active venous thromboembolic disorder (e.g. deep vein thrombosis, pulmonary embolism);
* A subject must not have a history or presence of severe hepatic disease with AST and/or ALT levels of >=3 times the upper normal limit;
* A subject must not have congenital or acquired malformations or distortions of the uterus or cervix;
* A subject must not have large or multiple uterine fibromyomata, or a smaller uterine fibromyoma which may interfere with the insertion of the MIUS/IUD according to the investigator;
* A subject must not have vaginal bleeding of undiagnosed etiology;
* A subject must not have dysmenorrhea interfering with daily activities or menorrhagia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome for the trial is insertion and removal characteristics, adverse event reporting and subject's satisfaction with the ENG-MIUS | 6 months

SECONDARY OUTCOMES:
Vaginal bleeding pattern | Days 92 to 182